CLINICAL TRIAL: NCT04698057
Title: Amoxicillin-clavulanate Alone or in Combination With Ciprofloxacin in Low-Risk Febrile Neutropenic Adult Patients: A Prospective, Double-blind, Randomized, Non-Inferiority Multicenter, Phase III Clinical Trial.
Acronym: ACACIA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No enrolment due to Covid-19
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACACIA
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Febrile Neutropenia
MeSH Terms: conditions — Febrile Neutropenia | interventions — Amoxicillin-Potassium Clavulanate Combination; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amoxicillin clavulanate + ciprofloxacin (Active Comparator): Treatment with amoxicillin-clavulanate 1g tib and ciprofloxacine 750mg bid for 5 days
  Interventions: Drug: Amoxicillin Clavulanate; Drug: Ciprofloxacin
- Amoxicillin clavulanate + Placebo (Experimental): Treatment with amoxicillin-clavulanate 1g tib for 5 days
  Interventions: Drug: Placebo; Drug: Amoxicillin Clavulanate

INTERVENTIONS:
Drug: Placebo — The aim of the study is to validate the desescalation of the treatment to stop ciprofloxacin prescription that may not impact the outcome of the patients but add toxicity and antibiotics selection. Placebo will be administred in the experimental arm
  Arms: Amoxicillin clavulanate + Placebo
Drug: Amoxicillin Clavulanate — Will be administred to all patients
Drug: Ciprofloxacin — Will be administred to patients in the standard of care arm
  Arms: Amoxicillin clavulanate + ciprofloxacin

SUMMARY:
In low risk neutropenic fever in cancer, standard of care is the association of amoxicillin clavulanate and ciprofloxacin. But in this population, the rate of fever related to infection is very low, leading to a overtreatment of the patients. The aim of this study is to validate a descalation of the antibiotherapy with safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Treated for a solid cancer or a hematological malignancy
* Presented with low-risk* febrile neutropenia due to chemotherapy with an expected duration of neutropenia ≤ 7 days
* Neutropenia is defined by an absolute neutrophil count ≤ 500/mm3.
* Fever is defined by temperature ≥ 38.3° or ≥ 38° twice during a 1-hour interval.
* Signing informed consent *Low risk is defined by MASCC score ≥ 21

Exclusion Criteria:

* Hypersensitivity to the active substances: amoxicillin-clavulanic, ciprofloxacin, penicillins, to other quinolones or to one of the excipient
* History of severe immediate hypersensitivity reaction to another beta-lactam
* History of jaunditis/hepatic impairment related to amoxicillin/clavulanic
* Concomitant administration of ciprofloxacin and tizanidine.
* Clinical signs of focal infection including history of untreated dental abscess.
* Signs of sepsis or organ failure.
* Severe immune deficiency other than the current cancer, except controlled-HIV infection
* Gastrointestinal symptoms requiring intravenous treatment (mucositis, vomiting, severe diarrhea...).
* Known aminotransferase serum levels > 5 x normal values.
* Known renal insufficiency defined as creatinine clearance of < 30 mL/min (MDRD).
* Antibiotherapy within 24h before enrollment. Prophylactic use of amoxicillin is an exclusion criterium whereas prophylactic use of trimethoprim-sulfamethoxazole (cotrimoxazole) and penicillin G (Oracilline®) are not and will be considered in the analysis.
* History of infection or colonization due to bacteria resistant to experimental drugs in the previous year
* Can be enrolled in the study only once.
* Patients not benefiting from a Social Security scheme or not benefiting from it through a third party.
* Persons benefiting from enhanced protection, namely minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection, and finally patients in emergencies
* Pregnant or breastfeeding women, women at age to procreate and not using effective contraception (either hormonal / mechanical : oral, injection, subcutaneous, implantable, intrauterine device, or surgical : tubal ligation, hysterectomy, total ovariectomy).

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Success rate | 7 days
  The success rate is defined by the proportion of patients receiving the tested regimen:
  * with resolution of fever ≤72h after the start of antibiotics (total duration of antibiotics expected : 5 days)
  * AND without any modification of the antibiotic regimen (route, dosage, combination total duration of antibiotics expected : 5 days),
  * AND without fever recurrence in 48h following the discontinuation of antibiotics (so end of the measure of the main outcome at day 7).